CLINICAL TRIAL: NCT05657626
Title: Examining of the Effect of Active Period Length of Firefighters on Respiratory Functions and Stair Climbing Performance
Brief Title: Effect of Active Period Length of Firefighters on Respiratory and Climbing
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: firefighters_study_1
Record Dates: First submitted 2022-12-09; First posted 2022-12-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-11

CONDITIONS: Firefighter; Respiratory; Climbing
Keywords: Firefighter; Respiratory; Climbing; Occupational exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cross-sectional study is to examine the effect of the active period of firefighters in the units on respiratory functions and stair climbing performance. In the relevant fire department, aged between 18 and 64, who do not have a psychological, cognitive or emotional problem, a chronic heart or lung disease that would prevent them from participating who have been active for at least two years, will be included.

The main questions it aims to answer are:

* What is the effect of the active period of firefighters on respiratory functions?
* What is the relationship between the length of active period of firefighters in the profession and their stair climbing performance?

Participants sociodemographic characteristics will be questioned by using the Demographic Data Form.

* Pulmonary function test and respiratory muscle strength measurement will be performed with the Pony Fx pulmonary function test device.
* The Cornell Musculoskeletal Disorders Questionnaire will be used to evaluate musculoskeletal disorders.
* The 6 Minute Walk Test will be performed to evaluate exercise capacity.
* Stair Climbing Test will be applied to evaluate stair climbing performance.

DETAILED DESCRIPTION:
Firefighters are occupational groups that work in difficult conditions both in their professional lives and during their education. These difficult conditions can lead to some negative situations on the physical and mental health of firefighters. Exposure of firefighters to smoke or chemicals during operation and training can be given as an example of their negative effects. Exposure to chemical substances also causes respiratory problems in people. The effect of the active period of firefighters on respiratory functions should be examined. This issue was emphasized while creating the study objectives. Physical performance is also extremely important for firefighters.

The assessment of physical performance will focus on training and stair climbing activity, which also provides a measure of endurance capacity in operation. In the study, the effect of the active period of firefighters on respiratory functions and stair climbing performance will be examined. In the evaluation of the effect of the active period in the profession, measurement, survey studies and some tests will be carried out in a group of volunteer firefighters. The data to be obtained from the research will be associated with the age groups of the firefighters participating in the study and the active period they spent in the profession. The effect of occupational exposure on respiratory functions and stair climbing performance will thus be determined.

Individuals who signed the Informed Consent Form will be included in the study in accordance with the inclusion and exclusion criteria from among the firefighters. The sociodemographic characteristics of the firefighters participating in the study will be questioned by using the Demographic Data Form. Pulmonary function test and respiratory muscle strength measurement will be performed with the Pony Fx pulmonary function test device. The Cornell Musculoskeletal Disorders Questionnaire will be used to evaluate musculoskeletal disorders. The 6 Minute Walk Test will be performed to evaluate exercise capacity. Stair Climbing Test will be applied to evaluate stair climbing performance.

In this study, the effect of the active period of firefighters on respiratory functions and stair climbing performance will be examined. Through the examination, its relationship with physical performance and endurance will be determined. According to the results, it is expected to determine preventive approaches to prevent problems that may occur due to the length of the active period. With this study, it is anticipated that the researchers will gain practical skills and experience related to the targeted methodologies. At the same time, it is among our goals to present the results of the study as a paper in national and international scientific congresses and to publish them as articles in scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer firefighters working in the relevant fire department, aged between 18 and 64, who do not have a psychological, cognitive and emotional problem, who do not have a chronic heart or lung disease that would prevent them from participating in our study, who have been active for at least two years, will be included in the study.

Demographic information of the individuals included in the study will be obtained and an Informed Voluntary Consent Form will be signed. Firefighters who do not give written consent to participation will not be included in the study.

Exclusion Criteria:

* Have been working in the organization for less than 2 years
* Having a chronic respiratory illness before starting to work in the institution
* Refusing to participate in the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteer firefighters working in the relevant fire department, aged between 18 and 64, who do not have a psychological, cognitive and emotional problem, who do not have a chronic heart or lung disease that would prevent them from participating in our study, who have been active for at least two years, will participate in the study.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Demographic Information | 10 minutes
  The sociodemographic data of the firefighters will be questioned using the "Demographic Data Form". With this form, firefighters' age, gender, height, weight, marital status, smoking and alcohol use, fire service start date and time on duty, department type and rank, estimated number of fires responded to, estimated number of toxic exposures, specific work-related exposures injuries or illnesses, type and severity of injury, body part affected, event at the time of injury (fire location, transportation, training), factors causing injury (equipment failure, lack of training, firefighter fatigue), and sleepy dyspnea and coughing spells will be questioned.
Respiratory Muscle Strength Measurement: | 15 minutes
  Maximum inspiratory pressure and maximum expiratory pressure (MIP/MEP) measurements will be made with the Pony Fx respiratory function tester. In the MIP measurement, the participant will complete a slow expiration to the remaining volume level during the test and make a rapid inspiration. The participant's inspiratory force will be measured using a pressure gauge against the closed shutter. Standard mouthpieces and nose clips will be used during the test. In MEP measurement; will be measured when the participant reaches the total lung volume level. In the meantime, the pressure created by the rapid expiration will be measured by the sensors. After 1.5-2.0 seconds the shutter will open and the test will end. In cases where more than one test is required, a maximum of 3-5 tests will be performed and the participant will rest for at least 1 minute between the two tests. The highest rating achieved will be recorded with the expected value.
Pulmonary Function Test | 15 minutes
  The test will be done with the Pony Fx pulmonary function tester. In order for the test to be administered, the participant will first be given the correct position. Then the nose clip will be attached, the mouthpiece will be placed and care will be taken to keep the lips closed. The participant will perform a rapid and deep inspiration, thereby reaching the total lung volume level. A strong expiration will then be requested without holding the breath for more than 1 second, and the maximal expiratory maneuver will be continued until the lungs are empty. Care will be taken not to perform the Valsalva maneuver during the test. Care will be taken to ensure that the participant makes a maximal inspiration, initiates the expiratory maneuver well, and performs an uninterrupted and effortless expiration. The test is repeated 8 times, but if a valid maneuver is still not achieved or the person detects fatigue, the test is stopped.
6 Minutes Walk Test | 6 minutes
  It is the gold standard for assessing exercise capacity. A straight corridor of 30 meters is required for the test. Before starting and at the end of the test, heart rate, blood pressure, oxygen saturation, dyspnea and fatigue will be evaluated using the Modified Borg Scale. It is convenient to use portable, battery-operated measuring devices to check oxygen saturation and heart rate during the test. Before the test starts, the person will be told about the test. The person will walk along the corridor in 6 minutes. The physiotherapist will calculate the distance walked by the number of laps the person has walked. When the time is up, the individual will be seated and the level of dyspnea and fatigue according to the oxygen saturation, heart rate, blood pressure, Modified Borg Scale will be questioned again and the measurements will be recorded. The modified Borg scale ranges from 0 to 10, with the value closer to 10 indicating worsening of symptoms. 0: none. 10: the most severe
Cornell Musculoskeletal Disorders Questionnaire | 15 minutes
  "Cornell Musculoskeletal Disorders Questionnaire" will be used. This survey; It was developed for the evaluation of musculoskeletal disorders in the Cornell University workforce population. It has Turkish validity and reliability. The test includes evaluations of 20 body parts on three scales of musculoskeletal disturbance frequency, severity, and interference with work capacity. While evaluating the frequency, it is questioned how many times he has felt the problem in the last week. Its severity is assessed as mild, moderate or very severe. The fact that the related musculoskeletal problem interferes with the workforce is also stated by the participant as none, a little and a lot. There are separate forms of the test for men and women. The risk score is obtained from the answers given and interpreted. Score, 1.5: mild discomfort. 1.6-10.5: moderate discomfort. Score >10.5: severe discomfort.
Stair Climbing Test | 15 minutes
  It will be applied to evaluate stair climbing performance. The test will be explained to the participants before it starts. Participants will be asked to go up and down the stairs once without wearing weighted vests to warm up. Participants will be given a command to start the test and they will be expected to go up and down the stairs without stopping 4 times, without holding on to the handrail or wall. Participants will be asked to touch each step with one foot as fast as possible, at the end of the fourth round, the time will be stopped when both feet touch the bottom court.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No